CLINICAL TRIAL: NCT05010980
Title: Early Detection of Cardiac Amyloidosis Among Patients With Aortic Valve Stenosis.
Brief Title: Early Detection of Cardiac Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 21-002
Record Dates: First submitted 2021-08-05; First posted 2021-08-18 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Amyloidosis; Aortic Valve Stenosis
Keywords: Amyloidosis; Aortic Valve Stenosis; MRI; myocardial scintigraphy; screening algorithm; early detection
MeSH Terms: conditions — Amyloidosis; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective: For the retrospective part of the study, the existing echocardiographic database will be used to retrieve data. The database query includes the last 2 years.
  Interventions: Other: CMR; Other: scintigraphy
- prospective: For the prospective part of the study, patients will be included who have the clinical indication for cmr and scintigraphy due to suspected cardiac amyloidosis and fulfill the inclusion criteria.
  Interventions: Other: CMR; Other: scintigraphy

INTERVENTIONS:
Other: CMR — clinical indication
Other: scintigraphy — clinical indication

SUMMARY:
Due to a lack of therapeutic options, the diagnosis of cardiac (wt)-ATTR amyloidosis was for a long time overshadowed by other diseases and therefore was or still is often diagnosed with considerable delay.

The aim of the study is to estimate the prevalence of cardiac amyloidosis among patients with mild-to-moderate aortic valve stenosis (AS).

Besides that a screening algorithm based on echocardiographic parameters will be developed, to facilitate the early detection of cardiac amyloidosis.

DETAILED DESCRIPTION:
Due to a lack of therapeutic options, the diagnosis of cardiac (wt)-ATTR amyloidosis was for a long time overshadowed by other diseases and therefore was or still is often diagnosed with considerable delay. On the one hand, it was assumed that the number of cases was significantly lower than the latest studies showed, and on the other hand, until the introduction of new therapeutic agents, there was no approved therapeutic option available, so that the corresponding diagnosis did not result in any therapeutic consequences.

This has changed fundamentally in recent years. For example, analyses of patients who underwent interventional aortic valve replacement (TAVI) as a result of high-grade AS demonstrated cardiac amyloidosis in up to 16% of these patients. Patients with (paradoxical) low flow low gradient (lflg) AS, which is echocardiographically characterized by a low stroke volume index (SVI), are particularly frequently affected. In light of these data, recent publications recommend the use of a low SVI, in conjunction with ECG criteria (low Sokolow-Lyon index) relative to echocardiographically determined left ventricular myocardial mass (SLI/ LVM) as a screening tool for the presence of amyloidosis in the patient population with high-grade aortic valve stenosis.

In patients with mild-to-moderate AS, the prevalence of amyloidosis and the validity of these methods has not yet been clarified. However, identification of these would be, of particular interest, especially in view of the new therapy options, since with the modern therapy methods can only improve prognosis if the diagnosis is made early.

When cardiac amyloidosis is suspected, three procedures are currently used in clinical practice

1. myocardial biopsy (BX)
2. cardiac MRI (CMR)
3. scintigraphy with 99mTc phosphates as tracer (scintigraphy)

Myocardial biopsy is not suitable as a broad screening method due to cost, effort, and limited feasibility at designated centers. It's rather a goldstandard for confirming nonconclusive findings or for further differential diagnosis or prognostic assessment.

Scintigraphy and CMR are the established and regularly used methods for the detection of cardiac amyloidosis.

Scintigraphy is a cost-effective examination that can be performed on an outpatient basis with low radiation exposure and high sensitivity and specificity for the detection of cardiac (ATTR) amyloidosis, especially in (still) asymptomatic patients. Scintigraphy is already recommended for the screening of ATTR amyloidosis. Besides scintigraphy, the CMR also offers good sensitivity (80%) and specificity (94%) for the diagnosis of cardiac amyloidosis, CMR also offers the advantage of a comprehensive cardiac differential diagnosis with possible exclusion of amyloidosis. It can also be performed on an outpatient basis, does not require a radiation-based procedure and can diagnose cardiac amyloidosis with high reproducibility, both with and without contrast medium. Which of the latter two examinations is more suitable for amyloidosis screening has not been conclusively determined. Although CMR and scintigraphy are regulary used for amyloidosis screening, it is not yet known, which of the two examinations is more suitable.

The aim of the study is to estimate the prevalence of cardiac amyloidosis in mild-to-moderate AS.

Furthermore, a screening algorithm based on echocardiographic parameters should be developed, to facilitate the early detection of cardiac amyloidosis: This would allow earlier initiation of therapy and thus better therapeutic success in patients with cardiac amyloidosis. Accordingly, a better quality of life as well as a prolonged survival of these severely affected patients could be expected Furthermore, the evaluation of follow-up investigation should clarify whether patients with cardiac amyloidosis suffer a faster progression of their AS than those without amyloidosis.

A comparison of the imaging modalities (CMR and SZG) will provide clues for further delineation of the indication. of these in order to develop targeted diagnostic algorithms that are as efficient as possible.

ELIGIBILITY:
Inclusion Criteria [retrospective/prospective]:

* Age > 65 years
* Patients who fulfill at least 3 of the following 4 criteria based on cardiac ultrasound examination, which results in the clinical indication for CMR and scintigraphy
* Evidence an aortic valve stenosis, defined as opening area according to velocity time integral (VTI) < 2cm2
* Hypertrophy of the interventricular septum (IVS) > 11mm
* Echocardiographically assesed reduced stroke volume index (SVI) (< 35 ml/m2)
* Reduced ratio of electrical signals of the heart (in the ECG) to the mass of the heart muscle (< 1.6 *10-2 mV/g/m2)

Exclusion Criteria:

* Patients who are incapable of giving consent,
* Age < 65 years
* patients who have not given their written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients undergoing a routine echocardiographic assessment which results in the clinical indication for CMR and scintigraphy among patients with aortic valve stenosis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
prevalence of cardiac amyloidosis in mild-to-moderate AS | up to two years
  estimating the prevalence of cardiac amyloidosis

SECONDARY OUTCOMES:
frequency of more rapid progression of AS in patients with cardiac amyloidosis than those without | up to two years
  frequency of more rapid progression of AS in patients with cardiac amyloidosis than those

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Westenfeld, MD, Principal Investigator — Division. of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Diseases and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided